CLINICAL TRIAL: NCT02151916
Title: Reducing Disease Burden and Health Inequalities Arising From Chronic Dental Disease Among Indigenous Children: an Early Childhood Caries Intervention
Brief Title: Preventing Early Childhood Caries in Indigenous Children: the Baby Teeth Talk Study
Acronym: BTT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Herenia P. Lawrence, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IDP-103988
Record Dates: First submitted 2014-05-27; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Dental Caries; Early Childhood Caries
Keywords: dental caries; early childhood caries; topical fluorides; fluoride varnish
MeSH Terms: conditions — Dental Caries | interventions — Dental Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dental care, AG, MI & fluoride varnish (Experimental): The intervention comprises four components; provision of dental care to the mother during pregnancy (2nd trimester), preventive treatment with fluoride varnish to the teeth of children, and two behavioral interventions, namely oral health anticipatory guidance and motivational interviewing with the caregiver/mother.
  Interventions: Other: Dental care, AG, MI & fluoride varnish
- Delayed intervention (Other): Three fluoride varnish applications to the teeth of children and oral health anticipatory guidance and motivational interviewing for the caregiver when the child is aged 24, 30 and 36 months. Dental care also will be offered to the mothers/caregivers in the delayed intervention group when their children are aged 2 to 3 years old. Before the children are aged 2 years, standard dental care will be the comparator, which usually involves provision of dental care only if the participant is in pain.
  Interventions: Other: Delayed intervention

INTERVENTIONS:
Other: Dental care, AG, MI & fluoride varnish — Dental care during pregnancy, or soon thereafter, will comprise of a screening oral examination, extractions, restorations, scaling and prophylaxis, if needed, and will take as many dental visits as required to achieve a non-diseased mouth. Fluoride varnish application to the teeth of children in the immediate intervention group will occur when children are aged 6 to 10 months (time of tooth eruption), 12 and 18 months, as well as at 24 months. Oral health anticipatory guidance and motivational interviewing for the caregivers/mothers in the immediate intervention group will occur during pregnancy and when the children are aged 6-10 months (time of tooth eruption), 12 and 18 months.
  Arms: Dental care, AG, MI & fluoride varnish
Other: Delayed intervention — Delayed intervention controlled design; all participants ultimately receive the benefits of the interventions. The intervention group receives the interventions when the mother is pregnant until the child is two years old. The delayed intervention group receives the interventions when the child is two years old until the child is three years old.
  Arms: Delayed intervention

SUMMARY:
The purpose of this study is to determine whether a combination of pre- and post-natal preventive and behavioral interventions is effective in preventing early childhood caries in Indigenous children.

Early childhood caries (ECC) causes profound suffering, frequently requiring expensive treatment under a general anesthetic. It is associated with other chronic childhood conditions such as otitis media and nutritional disorders, and is the strongest predictor of poor oral health in adulthood. Despite ECC being entirely preventable, marked ECC disparities exist between Indigenous and non-Indigenous children in Australia, New Zealand and Canada. If the burden of ECC and associated oral health inequalities experienced by Indigenous children in these nations are to be reduced, more needs to be done to ensure that appropriate preventive measures, together with support for maintaining optimal oral health, are provided to caregivers of such children in the early life stages. This will be an interventional study, with all participants receiving the intervention benefits. Pregnant Indigenous women residing in the three countries, their families and communities will be included. The intervention will be implemented from birth and continue for the first three years of a participating child's life. It will involve four components; dental care provided to the mother during pregnancy, fluoride varnish applications for the child, oral health anticipatory guidance and motivational interviewing. Following an Indigenous research framework and methodology, the intervention will be tailored at the individual- or family-level, with each caregiver or family progressing to the next level only when they are ready. Developing a culturally-appropriate ECC intervention that aims to improve child oral health, in full partnership with the Indigenous communities involved, will provide much needed evidence for policy makers to address the challenge of improved oral health and related outcomes for Indigenous children.

DETAILED DESCRIPTION:
The study seeks to determine whether the implementation of a culturally-appropriate early childhood caries intervention reduces dental disease burden and oral health inequalities among Indigenous children. The study is part of a tri-nation research project entitled "Reducing disease burden and health inequalities arising from chronic dental disease among Indigenous children: an early childhood caries intervention", being simultaneously conducted in Canada, Australia, and New Zealand. It was created in response to a Request for Applications for the International Collaborative Indigenous Health Research Partnership (ICIHRP) grant - a funding initiative of the Canadian Institutes of Health Research, the Health Research Council of New Zealand and the National Health and Medical Research Council of Australia.

The Baby Teeth Talk (BTT) Study, the Canadian arm of the project, is a community-based participatory research project being conducted in partnership with Aboriginal communities and organizations. BTT targets expectant mothers and their newborns, over a three-year intervention period. BTT has successfully recruited over 500 pregnant First Nations and Metis women living in urban and on-reserve communities in Ontario and Manitoba in the past two and a half years. This 5-year study promotes and offers good dental care during pregnancy and uses Motivational Interviewing (MI) and Anticipatory Guidance (AG) to counsel mothers on caring for their children's teeth. Presently, study participants have all given birth and fluoride varnish is being applied to their babies' teeth twice per year for 3 years by First Nations and non-First Nations community-based researchers associated with the project. At the same time, mothers continue to receive MI and AG in an effort to address the dietary and oral health concerns of their children. The goal of the study's multi-pronged approach is to intervene early enough in the child's life to prevent the onset of early childhood caries, or at least, reduce the rates of the disease to levels comparable to the general Canadian population so that fewer Indigenous children require dental treatment under general anesthesia.

The investigators have currently started the clinical oral examinations of the 2-year-old participants to assess the effectiveness of the investigators pre- and post-natal preventive and behavioral interventions to prevent caries in young Indigenous children. This is the point when the investigators collect the primary outcome data for the investigators project.

ELIGIBILITY:
Inclusion Criteria:

* Women who identify themselves as one of the Aboriginal Peoples in Canada (First Nations, Metis, Inuit) and/or who are pregnant with an Aboriginal child and live in the designated study areas.

Exclusion Criteria:

* Women who do not identify themselves as one of the Indigenous Peoples in Canada or are not pregnant with an Aboriginal child or do not live in the designated study areas.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Child dental caries incidence and increment, as measured by the dmft/s Indices | from birth to 2 years
  Child dental caries experience at age 2 years will be used to calculate the 2-year caries incidence and increment, as no child is born with dental caries.

SECONDARY OUTCOMES:
Caregiver oral health knowledge | from preconception to 3 years post-partum
  Assessed by comparing results from the caregiver baseline and 2- and 3-year follow-up questionnaires.
Caregiver oral self-care | from preconception to 3 years post-partum
  Assessed by comparing results from the caregiver baseline and 2- and 3-year follow-up questionnaires.
Caregiver dental service utilization | from preconception to 3 years post-partum
  Assessed by comparing results from the caregiver baseline and 2- and 3-year follow-up questionnaires.
Caregiver oral health-related self-efficacy | from preconception to 3 years post-partum
  Assessed by comparing results from the caregiver baseline and 2- and 3-year follow-up questionnaires.
Caregiver oral health literacy | from preconception to 3 years post-partum
  Assessed by comparing results from the caregiver baseline and 2- and 3-year follow-up questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Herenia P. Lawrence, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto Faculty of Dentistry, Toronto, Ontario, Canada